CLINICAL TRIAL: NCT04254107
Title: A Phase 1 Study of SEA-TGT (SGN-TGT) in Subjects With Advanced Malignancies
Brief Title: A Safety Study of SEA-TGT (SGN-TGT) in Advanced Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study closed due to portfolio prioritization
Sponsor: Seagen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SGNTGT-001; C5791001 (Other: Pfizer); 2019-004748-31 (EudraCT Number)
Record Dates: First submitted 2020-01-31; First posted 2020-02-05 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Non-small Cell Lung Cancer; Gastric Carcinoma; Gastroesophageal Junction Carcinoma; Classical Hodgkin Lymphoma; Diffuse Large B-cell Lymphoma; Peripheral T-cell Lymphoma; Cutaneous Melanoma; Head and Neck Squamous Cell Carcinoma; Bladder Cancer; Ovarian Cancer; Triple Negative Breast Cancer; Cervical Cancer
Keywords: NSCLC; cHL; HNSCC; TNBC; DLBCL; PTCL-NOS; Seattle Genetics
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Stomach Neoplasms; Lymphoma, Large B-Cell, Diffuse; Lymphoma, T-Cell, Peripheral; Melanoma; Squamous Cell Carcinoma of Head and Neck; Urinary Bladder Neoplasms; Ovarian Neoplasms; Triple Negative Breast Neoplasms; Uterine Cervical Neoplasms | interventions — Brentuximab Vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- SEA-TGT Monotherapy (Parts A and B) (Experimental): SEA-TGT
  Interventions: Drug: SEA-TGT
- SEA-TGT + sasanlimab Combination Therapy (Part C) (Experimental): SEA-TGT + sasanlimab
  Interventions: Drug: SEA-TGT; Drug: sasanlimab
- SEA-TGT + brentuximab vedotin Combination Therapy (Part D) (Experimental): SEA-TGT + brentuximab vedotin
  Interventions: Drug: SEA-TGT; Drug: brentuximab vedotin

INTERVENTIONS:
Drug: SEA-TGT — Given into the vein (IV; intravenously) on Day 1 of each 21-day cycle
  Other Names: SGN-TGT
Drug: sasanlimab — Given via injection under the skin (subcutaneous) on Day 1 of each 21-day cycle
  Arms: SEA-TGT + sasanlimab Combination Therapy (Part C)
Drug: brentuximab vedotin — Given by IV on Day 1 of each 21-day cycle
  Other Names: Adcetris
  Arms: SEA-TGT + brentuximab vedotin Combination Therapy (Part D)

SUMMARY:
This trial will look at a drug called SEA-TGT (also known as SGN-TGT) to find out whether it is safe for patients with solid tumors and lymphomas. It will study SEA-TGT to find out what its side effects are. A side effect is anything the drug does besides treating cancer. It will also study whether SEA-TGT works to treat solid tumors and lymphomas.

The study will have four parts. Part A of the study will find out how much SEA-TGT should be given to patients. Part B will use the dose found in Part A to find out how safe SEA-TGT is and if it works to treat solid tumors and lymphomas. Part C will study how well SEA-TGT with sasanlimab works to treat solid tumors. Part D will study how well SEA-TGT with brentuximab vedotin works to treat classical Hodgkin lymphoma (cHL).

ELIGIBILITY:
Monotherapy Inclusion Criteria (Parts A and B)

* Histologically- or cytologically-confirmed advanced or metastatic malignancy, defined as:

  * One of the following tumor types:

    * Unresectable locally-advanced or metastatic non-small cell lung cancer (NSCLC), gastric/gastroesophageal (GE) junction carcinoma, cutaneous melanoma, head and neck squamous cell carcinoma (HNSCC), bladder cancer, cervical cancer, ovarian cancer, or triple negative breast cancer (TNBC)
    * Lymphomas, including:

      * cHL
      * Diffuse large B-cell lymphoma (DLBCL)
      * Peripheral T-cell lymphoma, not otherwise specified (PTCL-NOS)
    * Lymphoma: Participants should have disease progression on or after treatment with standard therapies expected to provide benefit in the judgement of the investigator.

      * cHL: Participants must have received at least 3 prior systemic therapies. Participants should have had disease recurrence or progression following brentuximab vedotin therapy or have been ineligible to receive brentuximab vedotin. Participants who have not received autologous stem cell transplant (SCT) must have refused or been deemed ineligible. Participants should have received or not be eligible to have received an anti-PD-1 agent.
      * DLBCL: Participants must have received at least 2 prior systemic chemo-immunotherapy regimens, including an anti-CD20 agent and combination chemotherapy. Unless clinically contraindicated, participants should have had disease that has relapsed after or be refractory to intensive salvage chemotherapy, including autologous SCT.
      * PTCL-NOS: Participants must have had at least 1 prior systemic therapy. Participants must have received or have been ineligible to receive the combination of cyclophosphamide, doxorubicin, vincristine, and prednisone (CHOP) or CHOP-like therapy. Participants with CD30-positive disease must have received or be ineligible to receive brentuximab vedotin. Participants must have also received intensive salvage therapy (defined as combination chemotherapy ± autologous SCT) unless they refused or were deemed ineligible.
* Measurable disease defined as:

  * Solid tumors: Measurable disease according to RECIST V1.1
  * Lymphomas: Fluorodeoxyglucose (FDG)-avid disease by positron emission tomography (PET) and measurable disease of ≥15 mm in the greatest transverse diameter by computed tomography (CT) scan, as assessed by the site radiologist.
* A representative archival tumor tissue sample should be available as follows: Participants must provide archived tumor tissue, if available, from the most recent biopsy (less than or equal to [≤] 12 months from screening). If archived tissue is not available, a fresh baseline tumor biopsy will be requested for any participant enrolled in Part B whose tumors are considered accessible and appropriate in the opinion of the investigator.
* ECOG Performance Status score of 0 or 1

Combination Inclusion Criteria (Part C)

* ECOG Performance Status score of 0 or 1
* NSCLC: histological or cytological confirmed metastatic disease. Participants must have received no prior anti-PD-1/PD-L1 therapy allowed.
* HNSCC: histological or cytological confirmed metastatic disease. Participants must have received no prior exposure to anti-PD-1/PD-L1 therapy.
* Cutaneous Melanoma: histological or cytological confirmed metastatic disease. Participants must not have received anti-PD-1/PD-L1 targeted therapy.
* Measurable disease by CT or magnetic resonance imaging (MRI) as defined by RECIST V1.1
* Participants must provide archival tumor tissue from the most recent biopsy (≤12 months from screening). If archival tissue is not available, a fresh baseline tumor biopsy that has not been previously irradiated is required for any participant whose tumors are considered accessible and appropriate in the opinion of the investigator.

Combination Inclusion Criteria (Part D)

* Histologically- or cytologically-confirmed advanced stage cHL
* cHL patients that have failed standard of care for R/R disease including prior treatment with BV.
* FDG PET emission tomography avid and bidimensional measurable disease of at least 1.5 cm in longest axis as documented by radiographic technique
* ECOG performance status of ≤ 2
* Participants are required to have tumor tissue, if available, from the most recent biopsy (≤12 months from screening) prior to start of study treatment. If archival tissue is not available, a fresh screening tumor biopsy is required for any participant whose tumors are considered accessible and appropriate in the opinion of the investigator.

Monotherapy Exclusion Criteria (Parts A and B)

* History of another malignancy within 2 years before the first dose of study drug, or any evidence of residual disease from a previously diagnosed malignancy. Exceptions are malignancies with a negligible risk of metastasis or death.
* Chemotherapy, radiotherapy, biologics, and/or other antitumor treatment that has not been completed before the first dose of study drug within the timeframe as follows:

  * Chemotherapy, small molecule inhibitors, radiation, and/or other investigational anticancer agents (excluding investigational monoclonal antibodies): 2 weeks

    * Palliative radiotherapy (≤2 weeks of radiotherapy to non-central nervous system [CNS] disease): ≤7 days prior to start of SEA-TGT
  * Immune-checkpoint inhibitors: 4 weeks
  * Monoclonal antibodies, antibody-drug conjugates (ADC), or radioimmunoconjugates: 4 weeks (2 weeks with documented disease progression)
  * T-cell or other cell-based therapies: 12 weeks
* Known CNS metastases

  * Participants with a history of CNS metastases are allowed if they have undergone treatment for the CNS disease, symptoms have resolved, and steroids have been discontinued.
  * Leptomeningeal involvement by malignant disease is excluded regardless of prior treatment.
* Previous allogeneic stem cell transplant (SCT). Participants with prior autologous SCT may be eligible if they are >100 days from autologous SCT and fulfill all other inclusion criteria.
* Prior use of any anti-TIGIT mAb.
* Participants with a condition requiring systemic treatment with either corticosteroids (greater than [>]10 mg daily prednisone or equivalent) or other immunosuppressive medications within 14 days of enrollment. Inhaled or topical steroids and adrenal replacement steroid doses >10 mg daily prednisone or equivalents are permitted in the absence of active immune disease.
* Known hypersensitivity to any excipient contained in the drug formulation of SEA-TGT

Combination Exclusion Criteria (Part C)

* History of another malignancy within 2 years before the first dose of study drug, or any evidence of residual disease from a previously diagnosed malignancy. Exceptions are malignancies with a negligible risk of metastasis or death.
* Active, non-infectious pneumonitis, pulmonary fibrosis, or known history of immune mediated pneumonitis.
* Previous therapy with an anti-PD-1 or anti-PD-L1 inhibitor.
* Chemotherapy, radiotherapy, biologics, and/or other antitumor treatment that has not been completed before the first dose of study drug within the timeframe as follows:

  * Chemotherapy, small molecule inhibitors, radiation, and/or other investigational anticancer agents (excluding investigational monoclonal antibodies): 2 weeks

    * Palliative radiotherapy (≤2 weeks of radiotherapy to non-CNS disease): ≤7 days prior to start of SEA-TGT.
  * Immune-checkpoint inhibitors: 4 weeks
  * Monoclonal antibodies, ADC, or radioimmunoconjugates: 4 weeks (2 weeks with documented disease progression)
  * T-cell or other cell-based therapies: 12 weeks
* Known active CNS metastases.

  * Participants with a history of CNS metastases are allowed if they have undergone treatment for the CNS disease, symptoms have resolved, and steroids have been discontinued.
  * Leptomeningeal involvement by malignant disease is excluded regardless of prior treatment.
* Known hypersensitivity to any excipient contained in the drug formulation of SEA-TGT or sasanlimab
* Participants with active known or suspected autoimmune disease or significant autoimmune-related toxicity from prior immuno-oncology-based therapy (prior autoimmune colitis, pneumonitis, transaminitis); Participants with vitiligo, controlled type 1 diabetes mellitus, residual hypothyroidism requiring hormone replacement, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
* History of interstitial lung disease
* Participants with a condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone or equivalent) or other immunosuppressive medications within 14 days of enrollment. Inhaled or topical steroids and adrenal replacement steroid doses >10 mg daily prednisone or equivalents are permitted in the absence of active immune disease.
* Prior use of any anti-TIGIT mAb

Combination Exclusion Criteria (Part D)

* History of another malignancy within 2 years before the first dose of study drug, or any evidence of residual disease from a previously diagnosed malignancy. Exceptions are malignancies with a negligible risk of metastasis or death.
* Chemotherapy, radiotherapy, biologics, and/or other antitumor treatment that has not been completed before the first dose of study drug within the timeframe as follows:

  * Chemotherapy, small molecule inhibitors, radiation, and/or other investigational anticancer agents (excluding investigational monoclonal antibodies): 2 weeks

    * Palliative radiotherapy (≤2 weeks of radiotherapy to CNS disease): ≤7 days prior to start of SEA-TGT
  * Immune-checkpoint inhibitors: 4 weeks
  * Monoclonal antibodies, ADC (except brentuximab vedotin), or radioimmunoconjugates: 4 weeks (2 weeks with documented disease progression)
  * T-cell or other cell-based therapies: 12 weeks
* Known active CNS involvement by lymphoma
* Previous allogeneic SCT. Participants with prior autologous SCT may be eligible if they are >100 days from autologous SCT and fulfill all other inclusion criteria.
* Prior use of any anti-TIGIT mAb.
* Participants with a condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone or equivalent) or other immunosuppressive medications within 14 days of enrollment. Inhaled or topical steroids and adrenal replacement steroid doses >10 mg daily prednisone or equivalents are permitted in the absence of active immune disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2020-05-29 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) | Through 45-52 days following last dose of SEA-TGT; up to approximately 3 years
  An AE is any untoward medical occurrence in a subject or clinical investigational subject administered a medicinal product and which does not necessarily have a causal relationship with this treatment.
Number of participants with laboratory abnormalities by grade | Through 45-52 days following last dose of SEA-TGT; up to approximately 3 years
  To be summarized using descriptive statistics
Number of participants with a dose-limiting toxicity (DLT) at each dose level | Up to 21 days
  To be summarized using descriptive statistics

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to approximately 3 years
  Proportion of participants with complete response (CR) and partial response (PR) per the participant's specific tumor response criteria
Complete response (CR) rate | Up to approximately 3 years
  Proportion of participants with CR per the participant's specific tumor response criteria
Duration of objective response | Up to approximately 3 years
  Time from first response to the first documentation of disease progression or death due to any cause
Duration of CR | Up to approximately 3 years
  Time from start of the first documentation of CR to the first documentation of confirmed tumor progression or to death due to any cause, whichever comes first
Duration of progression-free survival | Up to approximately 3 years
  Time from first dose to the first documentation of disease progression or death due to any cause
Duration of overall survival | Up to approximately 3 years
  Time from start of study treatment to the date of death due to any cause
Area under the concentration-time curve (AUC) | Through 45-52 days following last dose of SEA-TGT; up to approximately 3 years
  To be summarized using descriptive statistics.
Time to maximum concentration (tmax) | Through 45-52 days following last dose of SEA-TGT; up to approximately 3 years
  To be summarized using descriptive statistics.
Maximum concentration (Cmax) | Through 45-52 days following last dose of SEA-TGT; up to approximately 3 years
  To be summarized using descriptive statistics.
Trough concentration (Ctrough) | Through 45-52 days following last dose of SEA-TGT; up to approximately 3 years
  To be summarized using descriptive statistics.
Number of participants with antidrug antibodies (ADA) | Through 45-52 days following last dose of SEA-TGT; up to approximately 3 years
  To be summarized using descriptive statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Andres Forero-Torres, MD, Study Director — Seagen Inc.
Locations (36):
- United States (26):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Arizona Oncology Associates, PC - HOPE, Tucson, Arizona
  - City of Hope, Duarte, California
  - California Research Institute, Los Angeles, California
  - University of California, San Francisco | HDFCCC - Hematopoietic Malignancies, San Francisco, California
  - Yale Cancer Center, New Haven, Connecticut
  - Johns Hopkins Medical Center, Baltimore, Maryland
  - Maryland Oncology Hematology, P.A., Rockville, Maryland
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Minnesota Oncology Hematology P.A., Minneapolis, Minnesota
  - Mayo Clinic Rochester, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Weill Cornell Medicine, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Wake Forest Baptist Medical Center / Wake Forest University, Winston-Salem, North Carolina
  - University of Cincinnati Cancer Institute, Cincinnati, Ohio
  - Providence Portland Medical Center, Portland, Oregon
  - University of Pittsburgh Medical Center (UPMC)/Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Oncology - Austin Midtown, Austin, Texas
  - Texas Oncology - Baylor Sammons Cancer Center, Dallas, Texas
  - MD Anderson Cancer Center / University of Texas, Houston, Texas
  - Texas Oncology - Northeast Texas, Tyler, Texas
  - Oncology and Hematology Assoc of SW VA DBA Blue Ridge Cancer Care, Blacksburg, Virginia
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
  - Carbone Cancer Center / University of Wisconsin, Madison, Wisconsin
- Canada (2):
  - University of Alberta / Cross Cancer Institute, Edmonton, Alberta
  - University Health Network, Princess Margaret Hospital, Toronto, Other
- Institut Gustave Roussy, Villejuif, Other, France
- Italy (2):
  - Istituto Europeo di Oncologia, Milan, Other
  - Policlinico Universitario Agostino Gemelli, Rome, Other
- Spain (3):
  - Hospital Universitari Vall d'Hebron, Barcelona, Other
  - L'Institut Catala d'Oncologia, L'Hospitalet de Llobregat, Other
  - HM Centro Integral Oncologico Clara Campal, Madrid, Other
- United Kingdom (2):
  - Sarah Cannon Research Institute UK, London, Other
  - The Royal Marsden Hospital (Surrey), Sutton, Other